CLINICAL TRIAL: NCT05670808
Title: "The Effect Of Subcutaneous Epinephrine Dosage On Blood Loss In Surgical Incision"
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Erum Naz, resident of plastic surgery and reconstruction, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: erumnaz1
Record Dates: First submitted 2022-09-16; First posted 2023-01-04 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2022-12

CONDITIONS: To Determine the Optimal Doses of Adrenaline in Preventing Blood Loos in Participants Undergoing Supraclavicular Flap Surgery
Keywords: Plastic reconstructive surgery, blood loss, epinephrine, supraclavicular flap
MeSH Terms: conditions — Hemorrhage | interventions — Epinephrine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Epinephrine 1:200,000 (Experimental): In this group participants will receive the epinephrine concentration of 1:200,000 in normal saline
  Interventions: Drug: Epinephrine injection
- Epinephrine 1:400,000 (Experimental): In this group participants will receive the epinephrine concentration of 1:400,000 in normal saline
  Interventions: Drug: Epinephrine injection
- Placebo (Placebo Comparator): In this group participants will receive only 10 ml of normal saline (control group)
  Interventions: Drug: Epinephrine injection

INTERVENTIONS:
Drug: Epinephrine injection — Different doses on epinephrine will be administered to study arms to observe its impact on blood loss

SUMMARY:
Several studies have attempted to calculate the ideal epinephrine concentration for vasoconstriction, however there has been little consensus. These experiments were carried out on animals, and the degree of vasoconstriction was measured using a variety of methods. Animal studies aren't always reliable since animal capillary density differs from human capillary density. Furthermore, because the density of capillaries in the head and neck is 30 to 40% higher than in other parts of the body, previous studies may not adequately reflect the ideal epinephrine concentration for this highly vascular location. As a result of this study, clinicians will be able to determine the appropriate dose of epinephrine to control intraoperative bleeding. This study aims to determine the effect of different doses of epinephrine on volume of bleeding in surgical incisions in participants undergoing supraclavicular flap surgery.

DETAILED DESCRIPTION:
INTRODUCTION The supraclavicular fasciocutaneous flap has recently been described for the repair of pharyngeal, oral cavity, parotid, lateral skull base, and cutaneous defects, among other head and neck deformities.The usage of this flap has been demonstrated to be well tolerated by patients, with low donor site morbidity and good recipient site viability.The supraclavicular flap is fairly thick, has a colour and texture similar to the head and neck area, and has a clear and consistent blood supply. The fap is easy to prepare, and the surgery takes only a few minutes. With the advancement of plastic surgery, the use of the supraclavicular flap is gaining popularity.

Bleeding is one of the most common problems in plastic surgery, and epinephrine injections have long been used to reduce blood loss. Bleeding during surgery can lead to issues such as a drop in haemoglobin, which may necessitate a blood transfusion. Perioperative blood transfusion was found to have an immunosuppressive impact, increasing the risk of infection after surgery. Blood transfusion or mandibular plate rebuilding was similarly associated with severe tissue ablation and a major surgical defect.

Various approaches, such as controlled hypotensive state surgery and infiltration of vasoconstrictive medicines, have been utilized to reduce the quantity of bleeding during the operation. All of these techniques have their own set of difficulties and adverse effects. Vasoconstrictive medications, particularly subcutaneous epinephrine, are now widely utilized to limit bleeding in cosmetic and reconstructive procedures.Due of its potential cardiac and local toxic consequences, ephinephrine has limitations. Arrhythmias, tachycardia, hypertension, and pulmonary edema are all cardiac toxicities that are exacerbated by the administration of hydrocarbon anaesthetics. Delay in healing, lower wound tensile strength, skin necrosis, and higher infection rates are all local toxic consequences.

Because these problems are dose-related, determining the minimum ephinephrine concentration required for adequate hemostasis during head and neck surgery involving supraclavicular flap would vastly improve its margin of safety. To the best of our knowledge, no research has been done on the effect of epinephrine on bleeding in participants undergoing supraventricular flap surgery. However, a study that looked at the impact of varying dosages of epinephrine on the level of vasoconstriction revealed that there were no significant differences in blood flow reduction between epinephrine concentrations of 1:100,000, 1:200,000, and 1:400,000. Epinephrine 1:800,000, on the other hand, caused substantially less vasoconstriction. To achieve optimal initial hemostasis while avoiding potential adverse effects, we recommend administering an epinephrine concentration of 1:200,000 or 1:400,000.

Objective:

1. To determine the effect of different doses of epinephrine on volume of bleeding in surgical incisions in participants undergoing supraclavicular flap surgery
2. To determine the optimal doses of adrenaline in preventing blood loos in participants undergoing supraclavicular flap surgery

Rationale:

Several studies have attempted to calculate the ideal epinephrine concentration for vasoconstriction, however there has been little consensus. 5-9 These experiments were carried out on animals, and the degree of vasoconstriction was measured using a variety of methods. Animal studies aren't always reliable since animal capillary density differs from human capillary density. Furthermore, because the density of capillaries in the head and neck is 30 to 40% higher than in other parts of the body, previous studies may not adequately reflect the ideal epinephrine concentration for this highly vascular location.

As a result of this study, clinicians will be able to determine the appropriate dose of epinephrine to control intraoperative bleeding.

Operational Definition:

Measurement of bleeding The amount Bleeding will be measured by two methods

1. By Volumetric method in suction bottle:

   Intraoperative blood loss will be measured by direct measuring the volume of blood in the suction bottle
2. By Gauze pieces. If gauze is used, it will be weighted before use and again after use when it has been soaked with blood, with the excess weight of the saturated gauze being quantified in milliliters of blood loss. All gauzes of same weight will be selected and digital weighting machine will be used.

Safety of different dosage will be monitor by

1.Heart Rate: Heart rate of patients will be monitor at base line and 5 min of administering of Adrenaline 2 Blood Pressure: BP will of patients will be monitor at base line and 5 min of administering of Adrenaline

MATERIAL AND METHODS:

STUDYDESIGN: Single blinded Randomized control trial

STUDYARMS:

Epinephrine 1:200,000: In this group participants will receive the epinephrine concentration of 1:200,000 in normal saline Epinephrine 1:400,000: In this group participants will receive the epinephrine concentration of 1:400,000 in normal saline Placebo: In this group participants will receive only 10 ml of normal saline (control group) SETTING: Study will be conducted in the plastic surgery department of DUHS

DURATION OF STUDY: Six months after ERC approval SAMPLE SIZE: Once ERC approval is received, sample size will be estimated after conducting a pilot study.

SAMPLING TECHNIQUE: Non-Probability consecutive sampling SELECTION CRITERIA

Inclusion criteria:

* Age≥ 18 years
* Patients who are undergoing supraclavicular flap surgery
* Patients wishing to be a part of study.
* Either gender

Exclusion criteria:

* Participants with cardio vascular diseases.
* Participants with collagen vascular diseases
* Participant who are on non-steroidal anti-inflammatory drugs, anticoagulants, or aspirin. .

DATA COLLECTION PROCEDURE:

Study will be commenced after CPSP and ERC approval. An informed consent will be taken from all the eligible patients. All the eligible patients will randomly be divided into three above mentioned groups. Participants will be randomized using a random number generator in excel. It will be single blinded study, Researcher will know the drug concentration but the participant will not know that what they will get in the study. At the time of enrolment the patient will be informed regarding the all interventional group of the studies and the probabilities of falling in any one treatment group at the time of taking inform consent. In two interventional groups of participants, ten milliliters of epinephrine in normal saline with doses of 1:200,000 and 1:400,000 will be given subcutaneously under the specified flaps before making the incision. Only 10 milliliters of normal saline will be used in the control group. 15 minutes after the injection, incisions will be created, and flaps will be released from the donor area using a dermatome. Bleeding will be measured for 5 minutes by Volumetric method (Intraoperative blood loss will be measured by direct measuring the volume of blood in the suction bottle).

A predesigned questionnaire will be used to gather information about the blood loss and epinephrine concentration. The participant heart rate, rhythm and blood pressure will be closely monitor during the procedure to avoid any adverse event.

DATA ANALYSIS PROCEDURE:

Data will be entered and analyzed using SPSS version 26.0. Mean ±SD or Median (IQR) will be computed for all the quantitative variables like age, height, weight, BMI, duration of surgery, total blood loss and pre and post HB levels, based on the assumptions of normality. Normality will be checked using Shapiro Wilk test for normality. Frequency and percentage will be computed for all the qualitative variables like gender, co-morbid, occupation, BMI categories, indication of supra clavicular flap, site of surgery and requirement of blood .Chi-square test /Fisher exact test will be applied as appropriate to assess significant association between the treatment group co-morbid, occupation and BMI categories and requirement of blood transfusion. One-way ANOVA /Kruskal-Wallis test will be applied as appropriate to assess significant differences in mean Blood loss, duration of surgery, pre and post-surgery Hb levels between the study group. Effect modifiers such as age, BMI category, indication of surgery, site of surgery will be controlled through stratification. Post-stratification Chi-square/Fisher-Exact test will be applied as appropriate. P-value<0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Age≥ 18 years
* Patients who are undergoing supraclavicular flap surgery
* Patients wishing to be a part of study.
* Either gender

Exclusion Criteria:

* • Participants with cardio vascular diseases.

  * Participants with collagen vascular diseases
  * Participant who are on non-steroidal anti-inflammatory drugs, anticoagulants, or aspirin. .

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
Blood loss | 5 minutes
  Intraoperative blood loss will be measured by direct measuring the volume of blood in the suction bottle

IPD SHARING:
Plan to Share IPD: No